CLINICAL TRIAL: NCT01172301
Title: Leucine-enriched Essential Amino Acid Intake to Optimize Protein Anabolism in Children With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 104738
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Cystic Fibrosis
Keywords: CF; protein metabolism; essential amino acid intake
MeSH Terms: conditions — Cystic Fibrosis | interventions — Excitatory Amino Acids; Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral EAA vs total AA supplement (Experimental)
  Interventions: Dietary Supplement: Essential amino acid intake + Leucine vs total AA supplement

INTERVENTIONS:
Dietary Supplement: Essential amino acid intake + Leucine vs total AA supplement — 7 g as bolus
  Other Names: 7 g EAA + 40% LEU

SUMMARY:
Malnutrition, including muscle wasting commonly occurs in children with cystic fibrosis (CF), negatively influencing their quality of life and survival. At the time of a diagnosis of CF, severe protein deficits can already be present. It is important to get CF children fed adequately to prevent that their condition becomes worse or that recovery takes longer. Oral supplementation trials showed that gains in lean body mass are difficult to achieve in CF unless specific metabolic abnormalities are targeted. However, the specific needs for certain food components are not clear yet in children that are ill. Therefore, more information is necessary on the need for protein and certain amino acids in children with CF. Previous studies support the concept of essential amino acids (EAA) as an anabolic stimulus in the young and elderly and in insulin resistant states. Until yet no information is present on the anabolic effects of EAA in CF.

It is therefore our hypothesis that a high-leucine essential amino acids mixture specifically designed to stimulate protein anabolism will target the metabolic alterations of pediatric subjects with CF. In the present proposal, the acute metabolic effects of this high leucine essential amino acids mixture will be examined in pediatric subjects with CF and compared to that of a regular balanced total mixture of essential and non-essential amino acids. The principal endpoints will be the extent of stimulation of whole body protein synthesis as this is the principal mechanism by which either amino acid or protein intake causes muscle anabolism, and the reduction in endogenous protein breakdown. Both endpoints will be assessed by isotope methodology which is thought to be the reference method.

DETAILED DESCRIPTION:
In this study, we will test the following hypothesis: A high-leucine essential amino acid mixture (dose of 6.7 g) will stimulate protein anabolism to a greater extent than a standard balanced mixture of total (essential and non-essential) amino acids in CF pediatric subjects. The principal endpoints will be the extent of stimulation of protein synthesis rate and the reduction in endogenous protein breakdown. The current project will provide information that will enable us to better understand the underlying metabolic mechanisms that regulate protein metabolism in pediatric subjects with CF.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who already have a diagnosis of CF based on universal diagnostic criteria.
2. Age 14 to 21 years at the time of enrollment
3. Under routine medical control at the CF center of ACH
4. Admitted to the ACH for treatment of pulmonary exacerbation of CF disease.
5. Improvement in lung function (FEV1) at the time of enrollment back to baseline values (as determined in the clinically stable pre-hospital period)
6. Central or peripheral venous line in place
7. No planned major changes or interventions in the treatment and care of the pediatric subject on Day -2 and -1 before discharge from the hospital.

Exclusion Criteria:

1. Established diagnosis of Diabetes Mellitus
2. Presence of fever within the last 3 days
3. Unstable metabolic diseases including liver (cirrhosis) or renal disease
4. Chronic respiratory failure with cor pulmonale
5. Use of long-term oral corticosteroids or short course of oral corticosteroids in the preceding month before enrollment
6. Any other condition according to the principle investigator or study physician would interfere with collecting study samples
7. Failure to give assent / informed consent

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Net whole body protein synthesis rate | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement

SECONDARY OUTCOMES:
Whole body collagen breakdown rate | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Urea turnover rate | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Arginine turnover rate | Up to 2 years
  Measured in postabsorptive state
Liver protein synthesis rate | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Resting Energy expenditure | Up to 2 years
  Measured in postabsorptive state
Insulin kinetics | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Amino acid kinetics | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Glucose kinetics | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Fat-free mass | Up to 2 years
  Characterization of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas EP Deutz, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Engelen MP, Com G, Deutz NE. Increased whole body hydroxyproline production as assessed by a new stable isotope technique is associated with hip and spine bone mineral loss in cystic fibrosis. Clin Nutr. 2014 Dec;33(6):1117-21. doi: 10.1016/j.clnu.2013.12.008. Epub 2013 Dec 29. PMID 24423745